CLINICAL TRIAL: NCT02853643
Title: A Phase 1, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Food-Effect in Healthy Volunteers
Brief Title: Single Ascending Dose Study to Evaluate Pharmacokinetics and Food-Effect in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASN002-102
Record Dates: First submitted 2016-07-28; First posted 2016-08-03 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — gusacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25 mg Dose (Experimental): Single dose of 25 mg ASN002
  Interventions: Drug: ASN002
- 50 mg Dose (Experimental): Single dose of 50 mg ASN002
  Interventions: Drug: ASN002
- 100 mg Food effect cross over (Experimental): 100 mg single dose under both fasted and fed conditions in a cross over fashion
  Interventions: Drug: ASN002

INTERVENTIONS:
Drug: ASN002 — Single dose study with food effect

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, and determine the blood levels (pharmacokinetics), in both a fed and fasted condition, of a single dose of ASN002. Healthy volunteers will be participants in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, non-smoking subjects.
2. Willing to use contraception throughout the duration of the study and for 90 days after the study.
3. Capable of consent.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

1. Any clinically significant abnormality, infection, exposure to infection, recent live virus vaccination, or abnormal laboratory test results found during medical screening.
2. History of alcohol or drug abuse, or a positive urine drug screen or breath alcohol test at screening.
3. History of allergic reactions to protein kinase inhibitors, or significant allergic reactions to any drug.
4. Positive pregnancy test at screening.
5. Clinically significant ECG abnormalities.
6. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
7. Use of medication other than topical products without significant systemic absorption:
8. Donation of plasma within 7 days prior to dosing, or significant blood loss within the past 56 days.
9. Subject is pregnant, or breast feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting adverse events during the study | Days 1-28
  Safety and tolerability will be determined by the number of subjects reporting adverse events during the study.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Days 1-6
  Calculate Area under the plasma concentration time curve (AUC) from time 0 to infinity after first dose. AUC from time 0 to the time of last measured concentration. AUC from time 0 to 24 hours.
Area under the plasma concentration versus time curve (AUC) under fed and fasted conditions | Days 1-6
  Calculate Area under the plasma concentration time curve (AUC) from time 0 to infinity after first dose. AUC from time 0 to the time of last measured concentration. AUC from time 0 to 24 hours.
Maximum Plasma Concentration of ASN002 | Days 1-6
  Calculate observed maximum plasma concentration after a dose and observed maximum plasma concentration at steady state. The time to reach the peak plasma concentration. The time to reach the peak plasma concentration at steady state.
Maximum Plasma Concentration of ASN002 under fed and fasted conditions | Days 1-6
  Calculate observed maximum plasma concentration after a dose and observed maximum plasma concentration at steady state. The time to reach the peak plasma concentration. The time to reach the peak plasma concentration at steady state.
Drug half life of ASN002 | Days 1-6
  Calculate terminal elimination rate constant and terminal half-life of ASN002
Drug half life of ASN002 under fed and fasted conditions | Days 1-6
  Calculate terminal elimination rate constant and terminal half-life of ASN002

CONTACTS AND LOCATIONS:
Overall Officials: David Wyatt, MD, Principal Investigator — InVentiv Health Clinical Research Services
Locations (1):
- InVentiv Health, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No